CLINICAL TRIAL: NCT07088016
Title: A Comparative Study Between Lumbar Epidural Analgesia Versus Local Infiltration Anesthesia Combined With Dexmedetomidine Intravenous Infusion in Endoscopic Lumbar Discectomy Surgeries: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Egyptian Center for Research and Regenerative Medicine (Other Government)
Responsible Party: Principal Investigator, Maha Salah, Dr, Egyptian Center for Research and Regenerative Medicine
Other Study IDs: 6/02-2025
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Epidural Analgesics for Comparison
Keywords: epidural; dexmedetomidine; microscopic lumber discectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dexmedetomidine group: loading of Dexmedetomidine was done at a dose of 1 mcg/ kg over 10 minutes followed by continuous infusion at a rate of 0.5 mcg/kg/hr , followed by infiltration of the skin with 2-3 ml of lidocaine hydrochloride 1 % first by the surgeon then an 18 -G needle will be introduced to anesthetize the trajectory with 8-10 ml lidocaine 1 %. After reaching the superior articular process, 2-3 ml of lidocaine 1 % was used to anesthetize the facet joint.
- Epidural group: The epidural insertion point was 2 segments upper than the surgical procedure, 10 ml of Bupivacaine 0.25% was injected in the epidural space to adjust the sensory level. The epidural catheter will be removed after 2 hours from the end of the operation

SUMMARY:
The goal of this observational study is to compare the effectiveness and patient satisfaction of local anesthesia combined with intravenous Dexmedetomidine versus epidural anesthesia in endoscopic lumbar discectomy surgeries

DETAILED DESCRIPTION:
In recent years, with the development of medical instruments, minimally invasive surgical methods for lumbar disc herniation became increasingly popular, such as percutaneous transforaminal endoscopic discectomy (PTED) PTED under local anesthesia (LA) is recommended in consideration of safety. Under LA, patients keep conscious during the procedure, and the surgeon can obtain feedback directly from the patients if the nerve is interfered. However, in clinical practice, we found that many patients couldn't tolerate the pain during operation especially when placing the working channel Dexmedetomidine, a highly selective alpha 2 adrenoreceptor agonist, has unique characteristics in providing sedation and analgesia. Due to its central sympatholytic action, DEX produces dose-dependent sedation, antinociception and anxiolysis, while decreasing intraoperative hypertension and tachycardia episodes Epidural anesthesia is another major method which can keep patients awake during surgery and the surgeons can check the function of the nerve from the maintained motor function of patients' lower limbs

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to II.
2. Aged 18 to 60 years.
3. Both sexes.
4. Patients with clinical and radiological evidence of soft disc herniation in a single lumber segment.

Exclusion Criteria:

1. Spinal malformation
2. Recurrent lumber disc herniation (LDH)
3. Multi segment LDH
4. Patients younger than 18 years or older than 60 years
5. Patients with hypersensitivity to one of the used drugs
6. Patients suffering of coagulopathy
7. Operation time more than 1 hour

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients are American Society of anesthesiologists' physical status (ASA) I to II aged 18 to 60 years of both sexes with clinical and radiological evidence of soft disc herniation in a single lumber segment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
we compare numerical rating pain score (NRS) between the two groups immediately at foraminal dilatation maneuver | from January 2021 to January 2024
  It refers to the common method used in healthcare where patients rate their pain on a scale from 0 to 10:
  0 = No pain 10 = Worst pain imaginable.

SECONDARY OUTCOMES:
Heart rate (H.R) | from January 2021 to January 2024
  We compare the heart rate ( by beats per minute) in the 2 groups every 10 minutes intraoperative
Mean arterial blood pressure (MABP) | from January 2021 to January 2024
  we compare mean arterial blood pressure between the 2 groups by millimeter of mercury (mmhg) every 10 minutes intraoperative
we compare Bromage scale in the two groups intraoperative during foraminal dilatation by the surgeon | from January 2021 to January 2024
  It is a clinical tool used to assess motor function in the lower limbs following epidural or spinal anesthesia (from 0 to 3) 0 means full movement (no motor blockage) 3 means complete motor block - unable to move feet, legs, or raise leg.

CONTACTS AND LOCATIONS:
Locations (1):
- International Medical Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
"IPD will not be shared due to concerns regarding participant privacy, confidentiality, and regulatory limitations. In addition, appropriate consent for data sharing may not have been obtained from participants at the time of enrollment